CLINICAL TRIAL: NCT05229770
Title: Effect of Fruit Smoothie Supplementation on Psychological Distress Among People With Substance Use Disorders Receiving Opioid Agonist Therapy: a Randomised Controlled Trial
Brief Title: Effect of Fruit Smoothie Supplementation on Psychological Distress Among People Receiving Opioid Agonist Therapy
Acronym: FruktBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government); Helse Vest (Other); University of Bergen (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 155386/REK-A
Record Dates: First submitted 2022-01-24; First posted 2022-02-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Substance-Related Disorders
Keywords: Fruit; Food Supplementations; Opiate Substitution Treatment; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants randomised to the intervention arm will receive a 250 ml fruit smoothie as diet supplement for 20 weeks in addition to the regular OAT clinic follow-up. The fruit smoothies will be marketed products including combinations of the following fruits: apple, pineapple, mango, bananas, orange, blueberries, passion fruit, coconut, lime, and blackcurrant. The participants will receive a mixture of different smoothie types with the option of removing alternatives based on preferences. Fruit smoothie products will come in plastic bottles and will be delivered directly to the participants on a weekly basis. Each participant will receive a total of seven smoothie bottles per week with an oral agreement with each participant to consume one of these per day. Delivery of fruit smoothie will generally be given in parallel with delivery of OAT medication.
Who Masked: Outcomes Assessor
Masking Description: Even though complete blinding is regarded as difficult and infeasible, patients will be informed of the follow-up they will receive but not on other follow-up alternatives that are used or the exact hypotheses for the study. Outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fruit smoothie (Experimental): Participants randomised to the intervention arm will receive a 250 ml fruit smoothie as diet supplement for 20 weeks in addition to the regular OAT clinic follow-up. The fruit smoothies will be marketed products including combinations of the following fruits: apple, pineapple, mango, bananas, orange, blueberries, passion fruit, coconut, lime, and blackcurrant. The participants will receive a mixture of different smoothie types with the option of removing alternatives based on preferences. Fruit smoothie products will come in plastic bottles and will be delivered directly to the participants on a weekly basis. Each participant will receive a total of seven smoothie bottles per week with an oral agreement with each participant to consume one of these per day. Delivery of fruit smoothie will generally be given in parallel with delivery of OAT medication.
  Interventions: Dietary Supplement: Fruit smoothie
- Standard (No Intervention): Participants randomised to standard treatment will receive regular OAT clinic follow-up without added supplementation.

INTERVENTIONS:
Dietary Supplement: Fruit smoothie — Participants randomised to the intervention arm will receive a 250 ml fruit smoothie as diet supplement for 20 weeks in addition to the regular OAT clinic follow-up. The fruit smoothies will be marketed products including combinations of the following fruits: apple, pineapple, mango, bananas, orange, blueberries, passion fruit, coconut, lime, and blackcurrant. The participants will receive a mixture of different smoothie types with the option of removing alternatives based on preferences. Fruit smoothie products will come in plastic bottles and will be delivered directly to the participants on a weekly basis. Each participant will receive a total of seven smoothie bottles per week with an oral agreement with each participant to consume one of these per day. Delivery of fruit smoothie will generally be given in parallel with delivery of OAT medication.
  Arms: Fruit smoothie

SUMMARY:
Background: People with substance use disorders generally have poor diets including limited intake of fruit and vegetables. Evidence shows substantial health benefits from increasing fruit and vegetable consumption on a variety of indicators and possibly also psychological distress. A pilot study has indicated that supplementation with fruit smoothie could be promising also among people receiving opioid agonist therapy (OAT) for opioid dependence. FruktBAR will compare the efficacy of fruit smoothie supplementation within the OAT clinics compared to standard treatment.

Study design: FruktBAR is a multicentre, randomised controlled trial. The trial will recruit approximately 230 patients receiving OAT in Bergen and Stavanger, Norway.

Intervention: The intervention involves daily supplementation with 250 ml fruit smoothie. The main endpoints are 16 weeks after intervention initiation. Participants will be included and followed up during and after intervention.

Study population: The target group will be patients with opioid dependence receiving OAT from involved outpatient clinics in Bergen and Stavanger.

Expected outcome: This study will inform on the relative advantages or disadvantages of a fruit supplementation in addition to the current medically and psychologically oriented treatment of people receiving opioid agonist therapy. If the supplementation is found to be safe and efficacious, it can be considered for further scale-up.

DETAILED DESCRIPTION:
See below each section

ELIGIBILITY:
Inclusion Criteria:

* Receiving OAT from an included outpatient clinic with outpatient follow-up on weekly basis
* Having fruit and vegetable intake below 3 portions per day (assessed at screening)
* Confirming interest in participating in diet intervention (criteria specified)
* Giving informed consent

Exclusion Criteria:

* Allergies or prior anaphylactic reactions involving fruits or vegetables
* Poorly regulated diabetes type 1 or 2 (HbA1c >60 mmol/mol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Psychological distress | Mid of the intervention period 16 weeks after initiation
  The primary outcome is psychological distress assessed with the Norwegian validated translation ten item version of Hopkins Symptom Checklist (SCL-10) in the mid of the intervention period 16 weeks after initiation (12-20). This will be evaluated with mean SCL-10 item score and compared between intervention and control arm.

SECONDARY OUTCOMES:
Biochemical indicator of inflammation | Mid of the intervention period 16 weeks after initiation
  Biochemical indicators of inflammation measured with C-reactive protein in serum
Biochemical indicators of fruit intake | Mid of the intervention period 16 weeks after initiation
  Biochemical indicators of fruit intake measured with serum carotenoids
Fatigue Symptom Scale | Mid of the intervention period 16 weeks after initiation
  Changes in fatigue will be assessed with the Fatigue Symptom Scale (FSS-3, scale 0-18, higher values is worse)
Physical functioning | Mid of the intervention period 16 weeks after initiation
  Physical functioning assessed with 4-minute step-test measuring number of steps climbed in period
Health-related quality of life | Mid of the intervention period 16 weeks after initiation
  Changes in health-related quality of life will be assessed with EuroQoL EQ-5D-5L (0-100, higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fadnes, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - LAR Helse Stavanger HF, Stavanger, Rogaland
  - Department of Addiction Medicine, Haukeland University Hospital, Bergen, Vestland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javadi Arjmand E, Thomassen LM, Druckrey-Fiskaaen KT, Furulund E, Vold JH, Madebo T, Blomhoff R, Daltveit JT, Henriksen HB, Chalabianloo F, Johansen KA, Lid TG, Fadnes LT; ATLAS4LAR study group. The effect of fruit smoothie supplementation on psychological distress and biomarkers among people with opioid dependence receiving opioid agonist therapy: a randomized controlled trial. BMC Med. 2025 Aug 29;23(1):505. doi: 10.1186/s12916-025-04347-w. PMID 40877839
- [Derived] Fadnes LT, Furulund E, Druckrey-Fiskaaen KT, Madebo T, Vold JH, Olsvold M, Pierron MC, Carlsen SL, Blomhoff R, Lid TG; ATLAS4LAR Study Group. Effect of fruit smoothie supplementation on psychological distress among people with substance use disorders receiving opioid agonist therapy: protocol for a randomised controlled trial (FruktBAR). BMC Nutr. 2022 Sep 3;8(1):97. doi: 10.1186/s40795-022-00582-z. PMID 36057629
- See also: Description of ATLAS4LAR — https://helse-bergen.no/avdelinger/rusmedisin/rusmedisin-seksjon-forsking/bar/atlas4lar-kartlegging-og-behandling-av-lungesykdom-i-legemiddelassistert-behandling